CLINICAL TRIAL: NCT03734263
Title: Pilot Clinical Trial to Investigate the Safety and Efficacy of Phenylbutyrate Therapy for Patients With Pyruvate Dehydrogenase Complex Deficiency.
Brief Title: Use of Phenylbutyrate Therapy for Patients With Pyruvate Dehydrogenase Complex Deficiency.
Acronym: TIGEM2-PDH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Telethon (Other)
Responsible Party: Principal Investigator, Nicola Brunetti-Pierri, Principal Investigator, Fondazione Telethon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIGEM2-PDH
Record Dates: First submitted 2018-10-25; First posted 2018-11-07 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Pyruvate Dehydrogenase Complex Deficiency
MeSH Terms: conditions — Pyruvate Dehydrogenase Complex Deficiency Disease | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Intervention Model Description: An open-label, uncontrolled, multicentric clinical trial will be performed on pediatric patients with PDC deficiency. Enrolled subjects will receive a four-week period of treatment with NaPB; primary and secondary endpoints will be evaluated at defined time points. Before NaPB treatment, all patients will undergo a four-week period of observation during which the same parameters will be analyzed at different time points, with the aim of evaluating basal conditions in the absence of treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label (Experimental): sodium phenylbutyrate
  Interventions: Drug: sodium phenylbutyrate

INTERVENTIONS:
Drug: sodium phenylbutyrate — Enrolled subjects will receive a four-week period of treatment with sodium phenylbutyrate (oral use)

SUMMARY:
In this study phenylbutyrate is used for patients with pyruvate dehydrogenase complex deficiency. The aim of the study is to investigate the safety and efficacy of therapy.

DETAILED DESCRIPTION:
The Investigator will evaluate the safety and efficacy of a 4-weeks treatment with sodium phenylbutyrate in patients with pyruvate dehydrogenase complex deficiency. Efficacy will be evaluated based on biochemical endpoints (blood lactate and pyruvate).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be older than 3 months old and younger than 18 years old.
2. Clinical diagnosis of PDC deficiency confirmed by DNA testing showing a missense mutation in the PDHA1 gene.
3. Lactate concentration ≥ 2.5 mmol/l or ≥ 2 mmol/l, respectively in venous or arterial blood samples.
4. Provision of signed and dated informed consent form by the parents/legal guardians of the patient
5. Negative pregnancy test for women of childbearing potential, and agree to use effective form of contraception until 6 weeks post treatment.

Exclusion Criteria:

1. Frameshift or nonsense mutations of the PDHA1 gene.
2. Defects affecting any gene encoding PDC subunits other than PDHA1
3. Secondary forms of lactic acidosis (e.g. impaired oxygenation or circulation).
4. Tracheostomy or requirement for artificial ventilation.
5. Hyperlactatemia or organic acidosis associated with other metabolic disorders (e.g. biotinidase deficiency, primary disorders of gluconeogenesis, organic acidurias, primary defects of fatty acids oxidation)
6. Evidence of hepatic insufficiency, renal insufficiency, edema with sodium retention, cardiac arrhythmia, congenital heart defects, hypertension, blood dyscrasia, symptomatic pancreatitis, or inflammatory bowel disease.
7. Any clinical condition or medications known to significantly affect renal clearance.
8. Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful completion of the study.
9. Known allergic reactions to components of the study agent.
10. Treatment with another investigational drug or other intervention (including DCA) or participation in a clinical study with an investigational drug within 6 months prior to enrolment.
11. Pregnancy or lactation.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Efficacy: blood lactate (mmol/L) | two weeks after starting therapy
  blood lactate (mmol/L)
Efficacy: blood lactate (mmol/L) | four weeks after starting therapy
  blood lactate (mmol/L)

SECONDARY OUTCOMES:
Efficacy: blood pyruvate (mmol/L) | two weeks after starting therapy
  blood pyruvate (mmol/L)
Efficacy:urinary lactate (mmol/mol crea) | two weeks after starting therapy
  urinary lactate (mmol/mol crea)
Efficacy: blood pyruvate (mmol/L) | four weeks after starting therapy
  blood pyruvate (mmol/L)
Efficacy: urinary lactate (mmol/mol crea) | four weeks after starting therapy
  urinary lactate (mmol/mol crea)
Safety and tolerability:Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | two weeks after starting therapy
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Safety and tolerability: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | four weeks after starting therapy
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Napoli, Italy

REFERENCES:
- [Background] Ferriero R, Manco G, Lamantea E, Nusco E, Ferrante MI, Sordino P, Stacpoole PW, Lee B, Zeviani M, Brunetti-Pierri N. Phenylbutyrate therapy for pyruvate dehydrogenase complex deficiency and lactic acidosis. Sci Transl Med. 2013 Mar 6;5(175):175ra31. doi: 10.1126/scitranslmed.3004986. PMID 23467562
- [Background] Ferriero R, Brunetti-Pierri N. Phenylbutyrate increases activity of pyruvate dehydrogenase complex. Oncotarget. 2013 Jun;4(6):804-5. doi: 10.18632/oncotarget.1000. No abstract available. PMID 23868807
- [Background] Ferriero R, Boutron A, Brivet M, Kerr D, Morava E, Rodenburg RJ, Bonafe L, Baumgartner MR, Anikster Y, Braverman NE, Brunetti-Pierri N. Phenylbutyrate increases pyruvate dehydrogenase complex activity in cells harboring a variety of defects. Ann Clin Transl Neurol. 2014 Jul;1(7):462-70. doi: 10.1002/acn3.73. Epub 2014 Jun 19. PMID 25356417
- [Background] Ferriero R, Iannuzzi C, Manco G, Brunetti-Pierri N. Differential inhibition of PDKs by phenylbutyrate and enhancement of pyruvate dehydrogenase complex activity by combination with dichloroacetate. J Inherit Metab Dis. 2015 Sep;38(5):895-904. doi: 10.1007/s10545-014-9808-2. Epub 2015 Jan 20. PMID 25601413